CLINICAL TRIAL: NCT00319306
Title: Real Life Effectiveness in Asthma of Symbicort Single Inhaler Therapy
Acronym: RELEASE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5890L00012; RELEASE
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Last update posted 2009-03-17 (Estimated); Status verified 2009-03

CONDITIONS: Asthma
Keywords: Respiratory Tract Diseases; Bronchial Diseases; Anti-asthmatic agents; Anti-asthmatic drugs; Bronchodilators
MeSH Terms: conditions — Asthma; Respiratory Tract Diseases; Bronchial Diseases | interventions — Budesonide, Formoterol Fumarate Drug Combination

INTERVENTIONS:
Drug: Budesonide/formoterol
Device: Symbicort® Turbohaler®

SUMMARY:
The purpose of this study is to determine whether patients with asthma are better able to manage and control their symptoms by using one inhaler daily that both prevents as well as treats the symptoms of an asthma exacerbation.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18
* Confirmed diagnosis of mild to moderate asthma by doctor
* Currently receiving inhaled corticoid-steroid medicine for treatment of asthma and requiring a review of current asthma treatment

Exclusion Criteria:

* Women who are pregnant, breast-feeding, or planning pregnancy
* Patients with a history of chronic obstructive pulmonary disease
* Patients using any beta blocker therapy
* Patients receiving steroid tablets or steroid injections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550
Dates: Start 2005-09; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
In a real life setting, to compare Symbicort® Single Inhaler Therapy with a patient's previous therapy (including low dose ICS), by assessment of the changes in the Asthma Control Questionnaire score in uncontrolled asthmatic patients.

SECONDARY OUTCOMES:
Change in forced expiratory volume in one second (FEV1)
Change in peak expiratory flow (PEF)
Patient Reported Outcomes: AQLQ(S), SATQ, RCP-3 scores

CONTACTS AND LOCATIONS:
Overall Officials: Iain Small, MD, Principal Investigator — General Practitioner; AstraZeneca UK Medical Director, MD, Study Director — AstraZeneca
Locations (59):
- United Kingdom (59):
  - Research Site, Fowey, Cornwall
  - Research Site, Hove, East Sussex
  - Research Site, Ilford, Essex
  - Research Site, Glenrothes, Fife
  - Research Site, Dartford, Kent
  - Research Site, Airdrie, Lanarkshire
  - Research Site, Hamilton, Lanarkshire
  - Research Site, Doncaster, North Yorkshire
  - Research Site, Cookstown, Northern Ireland
  - Research Site, Downpatrick, Northern Ireland
  - Research Site, Barry, South Glamorgan
  - Research Site, Chase Terrace, Staffordshire
  - Research Site, East Horsley, Surrey
  - Research Site, Crawley, West Sussex
  - Research Site, Box, Wiltshire
  - Research Site, Bradford-on-Avon, Wiltshire
  - Research Site, Ashford
  - Research Site, Atherstone
  - Research Site, Ayrshire
  - Research Site, Bath
  - Research Site, Blackpool
  - Research Site, Bolton
  - Research Site, Cardiff
  - Research Site, Carrickfergus
  - Research Site, Cheshire
  - Research Site, Chesterfield
  - Research Site, Coventry
  - Research Site, Dundee
  - Research Site, Ellesmere Port
  - Research Site, Fife
  - Research Site, Glasgow
  - Research Site, Harrow
  - Research Site, Larne
  - Research Site, Leeds
  - Research Site, Middlesbrough
  - Research Site, Newcastle
  - Research Site, Newtownabbey
  - Research Site, Peterhead
  - Research Site, Pontypridd
  - Research Site, Reading
  - Research Site, Rugby
  - Research Site, Rutherglen
  - Research Site, Sandy
  - Research Site, Sheffield
  - Research Site, Stafford
  - Research Site, Stevenage
  - Research Site, Stockport
  - Research Site, Sunbury-on-Thames
  - Research Site, Sutton Coldfield
  - Research Site, Tilehurst
  - Research Site, Tonbridge
  - Research Site, Trowbridge
  - Research Site, Vale of Glamorgan
  - Research Site, Warminster
  - Research Site, Watford
  - Research Site, Wells-next-the-Sea
  - Research Site, Westbury
  - Research Site, Woking
  - Research Site, Yaxley